CLINICAL TRIAL: NCT00555555
Title: A Post-marketing Observational Study to Assess the Efficacy and Safety of the FVIII/VWF Complex (Human), Alphanate®, in Preventing Excessive Bleeding During Surgery in Subjects With Congenital Type 3 Von Willebrand Disease
Brief Title: Efficacy of Alphanate FVIII/VWF Concentrate in Type 3 Von Willebrand Patients
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Grifols Biologicals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBI 07-03
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Von Willebrand Disease
Keywords: Factor VIII deficiency; Von Willebrand disease; FVIII/VWF concentrate; Bleeding disorders; Blood disorders
MeSH Terms: conditions — von Willebrand Diseases; Hemophilia A; Hemostatic Disorders; Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Coagulation FVIII/VWF (Experimental): Anti-Hemophilic/von Willebrand Factor VIII (Human) Alphanate SD/HT
  Interventions: Biological: Alphanate SD/HT

INTERVENTIONS:
Biological: Alphanate SD/HT — A general guideline based on the product Full Prescribing Information is recommended with a maximum dose of 80 VWF:RCof IU/kg. The number of administrations before, during, and after the surgery procedure depends on the subject's clinical condition and the type of surgery itself. Single administrations or multiple doses may be appropriate. The dose of Alphanate® administered to each subject will be recorded as IU of VWF:RCof and also as IU of FVIII:C. The lot number for each vial of concentrate administered will also be recorded.
  Other Names: Alphanate® Factor VIII/VWF concentrate (Human)

SUMMARY:
To assess the efficacy of FVIII/VWF Complex (Human), Alphanate® as replacement therapy in preventing excessive bleeding in subjects with congenital Type 3 von Willebrand Disease (VWD) who undergo surgical procedures.

DETAILED DESCRIPTION:
For the treatment of surgical procedures the intended dose of Alphanate® will be given as a single dose or as multiple doses over several days, depending on the clinical situation, and according to the Full Prescribing Information guideline and the investigator's judgment. For each treated event, the subject's treatment period will be finished when, in the opinion of the local Investigator, the participating subject would not benefit from further infusions of the study concentrate.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 7 years of age or older
2. The subject has been diagnosed of inherited VWD of Type 3 as determined by subject's medical records.
3. The subject needs a surgical procedure (at least 10 surgical procedures have to be considered as "Major" according to the criteria of the protocol).
4. The subject is expected to respond to exogenously administered FVIII/VWF according to Investigator's judgment.
5. The subject freely gives written informed consent. Patients who are not legally permitted to provide written consent must sign a form of assent for study participation, and written consent must be provided by a parent or legal guardian.

Exclusion Criteria:

1. The subject has been diagnosed of acquired VWD.
2. The subject is known to have history of intolerance to any Alphanate® containing substance.
3. The subject is known to have history of anaphylactic reaction(s) to blood or blood components.
4. Liver function tests (AST, ALT, bilirubin) > 2.5 x upper limit of normal (ULN).
5. Renal function test (creatinine, BUN) > 1.5 x ULN.
6. The subject is known or suspected to have present or past inhibitor activity (antibodies) directed against FVIII or VWF.
7. The subject is known to abuse alcohol or illicit drug use within the past 12 months.
8. The subject is participating in another clinical study involving an investigational treatment, or participated within the past 4 weeks (except if the patient is participating in another Alphanate® study). Studies consisting of data and blood sampling collections on a regular or long-term basis are exempt from this exclusion.
9. The subject is unlikely to adhere to the protocol requirements of the study.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2007-09 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Assess the efficacy of FVIII/VWF Complex (Human), Alphanate® as replacement therapy in preventing excessive bleeding in subjects with congenital Type 3 von Willebrand Disease (VWD) who undergo surgical procedures (mostly major surgeries). | 30 days

SECONDARY OUTCOMES:
To assess the Day 0 (surgery day) and Day 1 (post-surgery day) treatment outcomes of each surgical procedure, rated by the investigator using a 2-point verbal rating scale. | 1 Day
Assessment of Safety and Tolerability | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Pinciaro, PhD, Study Director — Grifols Biologicals, LLC

IPD SHARING:
Plan to Share IPD: No